CLINICAL TRIAL: NCT01902810
Title: Protective Effects of Propranolol in Adults Following Major Burn Injury: A Safety and Efficacy Trial
Brief Title: Protective Effects of Propranolol in Adults
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: At the request of the study site, this study has been closed and access to study-related data is unavailable. We are unable to submit the results-data.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); American Burn Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-205
Record Dates: First submitted 2013-06-24; First posted 2013-07-18 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2018-08

CONDITIONS: Burn
MeSH Terms: conditions — Burns | interventions — Propranolol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propranolol (Active Comparator): Propranolol by mouth given daily throughout hospitalization
  Interventions: Drug: Propranolol
- Sugar Pill (Placebo Comparator): Placebo by mouth given daily throughout hospitalization
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Propranolol by mouth given daily throughout hospitalization
  Other Names: metoprolol; inderol
  Arms: Propranolol
Drug: Placebo — Placebo by mouth given daily throughout hospitalization
  Other Names: control
  Arms: Sugar Pill

SUMMARY:
This efficacy and safety trial will examine the effects and safety of propranolol administered to adult patients with severe burn injury. The investigators hypothesize that propranolol will provide significant benefit to adults following severe burn injury at doses that are safe and do not increase risk of adverse infectious and non-infectious outcomes.

DETAILED DESCRIPTION:
A safety and efficacy trial is needed in order to determine the safety of propranolol treatment in adult burn patients, identify which subpopulations may be most likely to benefit from propranolol treatment and to identify propranolol dose levels that are not only safe but potentially effective.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 20% Total Body Surface Area (TBSA) burn with anticipated operation need on admission
* Age ≥ 18 years
* Admission within 72 hours of injury

Exclusion Criteria:

* Age <18
* Patients unlikely to survive injury or with ;age = total burn size ≥ 130
* Electrical or deep chemical burn
* Malignancy currently undergoing treatment or history of cancer treatment within 5 years
* History of HIV or AIDS
* Presence of anoxic brain injury that is not expected to result in complete recovery
* Currently treated for Chronic Obstructive Pulmonary Disease (COPD), asthma or other chronic pulmonary conditions
* History of Congestive Heart Failure (CHF) (ejection fraction < 20%)
* Pre-injury medications including blocking agents (alpha or beta) or other anti-arrhythmic drugs
* Pregnant women
* Prisoners
* History of cardiac arrhythmia requiring medication
* Medical condition requiring glucocorticoid treatment
* Patients with concurrent conditions that in the opinion of the investigator may compromise patient safety or study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Cardiac rate pressure product | participants will be followed for the duration of hospital stay, an expected average of 5 weeks
  Multiply the subjects resting heart rate and blood pressure measurements as the average per 24 hours

SECONDARY OUTCOMES:
Mortality rates | time of randomization up to one year
  mortality rates will be compared between placebo group and propranolol treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Principal Investigator — University of Texas
Locations (10):
- United States (9):
  - University of Florida, Gainesville, Florida
  - Loyola University Burn Center, Maywood, Illinois
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Cornell Burn Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - University of Texas, Southwestern, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Washington, Seattle, Washington
- University of Toronto, Toronto, Ontario, Canada